CLINICAL TRIAL: NCT04524481
Title: Osteoporosis Screening in Adult Patients With Haemophilia and Influence of Physical Activity on the Prevalence of Osteoporosis
Brief Title: Osteoporosis and Haemophilia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PD Dr. Andreas Strauß (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. Andreas Strauß, specialist for orthopaedics and trauma surgery, University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Other Study IDs: NISOSTEO20200529; 2020-003072-41 (EudraCT Number)
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Osteoporosis; Haemophilia; Bone Mass
MeSH Terms: conditions — Osteoporosis; Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with mild haemophilia A or B: (FVIII or IX >5 %, ≥ 18 years' old)
- Patients with moderate haemophilia A or B: (FVIII or IX 1-5 %, ≥ 18 years' old)
- Patients with severe haemophilia A or B: (FVIII or IX <1 %, ≥ 18 years' old)

SUMMARY:
The aim of this study is to evaluate the prevalence of osteoporosis in adult patients with haemophilia.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the prevalence of osteoporosis in adult patients with haemophilia. Subsequently, the ascertained prevalence of osteoporosis in patients with haemophilia will be compared to the latest published data of osteoporosis in Germany. Furthermore, the impact of severity of haemophilia, comorbidities as well as the role of both physical activity and individual joint condition as influencing factors on the presence of osteoporosis will be analysed by this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) suffering from mild (FVIII or IX >5 %), moderate (FVIII or IX 1-5 %) or severe (FVIII or IX <1 %) haemophilia A or B
* Submitted written consent to participate in the study

Exclusion Criteria:

* Patients suffering from other bleeding diseases
* PWH without written consent
* PWH < 18 years of age
* Secondary osteoporosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) suffering from mild (FVIII or IX >5 %), moderate (FVIII or IX 1-5 %) or severe (FVIII or IX <1 %) haemophilia A or B
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
bone mass/bone density maesurement | 15 minutes
  All patients with haemophilia of this study will receive a standardised bone density measurement by using the same dual energy X-ray absorptiometry (DXA) device.
blood sample (Vit. D/Calcium) | 10 minutes
  The blood samples of all patients with haemophilia will be tested according to the guidelines of the confederation of osteology (DVO). These blood samples are necessary to assess the osteoporosis by measuring the Vitamin-D and Calcium level.

SECONDARY OUTCOMES:
haemophilia related clinical data | 10 minutes
  All patients with haemophilia record their individual substitution regime and bleeding events in individual patients' diaries. The patients are used to record and submit all necessary information about bleeding events, factor replacement regime. By doing so, the individual treatment regime per week as well as the annual (joint) bleeding rate will be assessed one year retrospectively.
level of physical activity | non determinable
  In order to assess the individual level of physical activity, an individual movement profile will be created. For this purpose, the activity of each patient with haemophilia will be recorded by an electronic activity tracker. In addition, the grade of individual physical activity will be assessed on the basis of questionnaires.
orthopaedic joint status | 45 minutes
  The clinical joint status will be examined in all patients with haemophilia by the World Federation Joint Examination Score and Haemophilia Joint Health Score.
pain condition | 15 minutes
  The pain condition will be examined in terms of pressure pain thresholds. By using an algometer device (Wagner Instruments, USA) with a robe area of 1 cm2 the individual pain sensitivity will be measured.
subjective quality of life and subjective physical performance | 10 minutes
  The examination of these parameters is carried out by the standardised questionnaires SF-36 (quality of life) and the HEP-Test-Q (subjective physical performance).

OTHER OUTCOMES:
blood samples | non determinable
  Blood samples of all PWH will be tested according to the guidelines of the confederation of osteology (DVO). Additionally, the liver's (GGT, GPT, GOT) and parathyroid glands' (PTH) function will be assessed and patient's will also be tested for testosterone-deficiency (testosterone), diabetes (HbA1c) and multiple myeloma (paracentesis).
  Furthermore these blood samples are necessary to define the immune phenotype (including: soluble mediators such as cytokines and growth factors, as well as the cellular immune composition, immune cell subsets and their detailed phenotype) to examine a possible correlation with the severity of osteoporosis.
Medical history | 10 minutes
  Medical history and pharmacological treatment will be recorded. Based on these parameters the occurrence of secondary osteoporosis will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Strauß, PD Dr., Principal Investigator — Medicine of the University of Bonn
Locations (1):
- University Hospital of Bonn, Bonn, Northrhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No
The publication of anonymous patient data is not allowed by informed consent.

REFERENCES:
- [Derived] Ransmann P, Bruhl M, Hmida J, Goldmann G, Oldenburg J, Schildberg FA, Ossendorff R, Tomschi F, Schmidt A, Hilberg T, Strauss AC. Physical activity and handgrip strength in patients with mild, moderate and severe haemophilia: Impacts on bone quality and lean mass. PLoS One. 2025 Mar 26;20(3):e0319951. doi: 10.1371/journal.pone.0319951. eCollection 2025. PMID 40138293